CLINICAL TRIAL: NCT00154895
Title: Phase III Study of Additional Minocycline Pleurodesis After Video-Assisted Thoracoscopic Surgery for Primary Spontaneous Pneumothorax
Brief Title: Additional Minocycline Pleurodesis After Thoracoscopic Procedures for Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 921204
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2001-06

CONDITIONS: Pneumothorax
Keywords: minocycline; pleurodesis; thoracoscopy; primary spontaneous pneumothorax; clinical trial
MeSH Terms: conditions — Pneumothorax; cyclopia sequence

INTERVENTIONS:
Drug: intrapleural minocycline instillation

SUMMARY:
To test if additional minocycline pleurodesis after thoracoscopic procedures can reduce the rates of ipsilateral recurrence for patients with primary spontaneous pneumothorax.

DETAILED DESCRIPTION:
Patients and Methods Study design This study is a randomized trial of additional minocycline pleurodesis after VATS for primary spontaneous pneumothorax. It was begun in June 2001 in Thoracic Surgical Division, National Taiwan University Hospital. After VATS for primary spontaneous pneumothorax, eligible patients were randomly assigned to additional minocycline pleurodesis or observation. The primary end point was rate of ipsilateral recurrence after the operation. Secondary end points included safety, early postoperative results, and long-term effects of minocycline pleurodesis. Consents were obtained from patients after thorough explanation. The protocol was approved by the Institutional Review Board of National Taiwan University Hospital.

Eligibility criteria All patients requiring VATS caused by ipsilateral recurrence, continuous air leaks for > 3 days, contralateral recurrence, presence of hemopneumothorax, or uncomplicated first episode with professions at risk were eligible for this study. The exclusion criteria were: greater than 50 years of age, underlying pulmonary disease, previous ipsilateral thoracic operation, allergy to tetracycline or minocycline, and unwillingness to randomization.

Operative technique of VATS After confirmation of patient eligibility, either conventional or needlescopic VATS was performed for these patients by his or her own choice. The cost of the operation and cosmetic results were the main points considered by the patients as they made their choices. The cost of needlescopic VATS is higher than that of conventional VATS because our National Health Insurance will cover only a part of the disposable equipment. Our previous study showed that the short-term results and recurrence rates of both techniques were comparable, although needlescopic VATS provides better cosmetic results and less residual chest pain.19 Conventional VATS was performed in a standard fashion under general anesthesia using intubation with a double-lumen endotracheal tube. The patients were placed in a lateral decubitus position, and the ipsilateral lung was deflated. A 10-mm, 30-degree telescope (Karl Storz, Tuttlingen, Germany) was first inserted to examine the pleural cavity. Two 15-mm skin incisions were made at the third or fourth intercostal space, anterior and posterior axillary line. Light pleural adhesions were freed using electrocautery. When blebs were identified, they were grasped with the ring forceps and excised with a 45-mm endoscopic stapler. Blind apical stapling was done at the most suspicious area if no bleb could be identified. The entire parietal surface was abraded by inserting the dissector with a strip of diathermy scratch pad through the port sites. After postoperative lung reinflation, normal saline solution was instilled to check for air leaks. A chest tube (28F) was placed in the apex through one of the insertion wounds. The surgical specimens were routinely sent for pathological examination.

The anesthesia, preparation, and operative procedures of the needlescopic VATS were almost identical to the conventional VATS. However, two sets of independent video-thoracoscopic equipment and monitors, one for needlescopic videothoracoscopy and the other for 10-mm videothoracoscopy, were used simultaneously and placed near the patient's head. Basically, we used the 10-mm videothoracoscopy for most of the surgical steps. A needlescope was indicated only when we need the chest tube wound to insert the endoscopic stapler and ring forceps, to extract the specimen, or to perform pleural abrasion.19

Postoperative care and minocycline pleurodesis The patients were extubated in the operating theater and observed for 1 to 2 hours in the recovery room. Postoperative analgesics include routine oral, non-steroid analgesics and acetaminophen. Intensity of postoperative pain was evaluated by a visual analogue scale (VAS; zero represented no pain and 10 represented intractable pain) on the first, second, and third postoperative days. Intramuscular meperidine hydrochloride (Demerol®, 50mg/ampule) was administered every 4 to 6 hours according to the patient's request if the pain became intolerable, could not be relieved by oral analgesics, and visual analogue scale was greater than 7. Chest radiography was performed immediate postoperatively or the next morning. The chest tube was connected to a low-pressure suction system of around -10 to -20 cmH2O if the lung was not fully expanded.

Randomization and treatment regimen Patients were randomized to additional minocycline pleurodesis (minocycline group) or observation (observation group) when the lung was expanded. Randomization was accomplished according to the chart number, which was randomly assigned before any kind of workup and management. When the chart number was even, the patient was allocated in the minocycline group. When the chart number was odd, the patient was allocated in the observation group. In the minocycline group, 20 mL of 2% lidocaine hydrochloride (400mg) followed by a solution of 20 mL of normal saline containing 300 or 400 mg (7mg/kg) of minocycline (Mirocin®, Taiwan Panbiotic Laboratories, Kaohsiung, Taiwan) was instilled into the pleural cavity through the thoracostomy tube. The rubber tube connecting the chest tube and chest bottle was raised 40 to 60 cm above the patient to trap the minocycline but allow air to pass under pressure. Patients were repositioned every 30 minutes so that the minocycline could contact all pleural surfaces. Side effects and complaints of the patient were recorded. The rubber tube was lowered 6 to 8 hours later.

To optimize the effects of pleural symphysis, minocycline was administered after full expansion of the lung, which was usually accomplished on the first postoperative day. However, in those patients who had persistent air leaks and could not fully inflate their lung, minocycline was still used after 3 to 5 days of waiting. In the observation group, nothing was instilled. A blinded study conducted by saline instillation was not suitable in our experiment because the pain associated with minocycline injection would unmask the blinding; and use of saline injection would place the patient at an unnecessary risk of contamination of the pleural space. When prolonged air leaks developed in the observation group, patients can still undergo minocycline instillation although the analysis was based on an intent-to-treat method. The tube was removed in both groups when the lung was fully expanded and no air leaks were noted in a 24-hour period.

All complications after the operation were recorded. Prolonged air leaks were defined when air leaks last for longer than 5 days. Pleural detachment was defined when a pneumothorax developed right after removal of the chest tube.

Follow-up After discharge from the hospital, patients were followed at the outpatient clinics at 1 week, 1 month, 3 months, and 6 months where chest radiography was performed. Follow-ups were then conducted every 6 months by a registered nurse who was blinded to the group allocation by telephone conversation, according to a standard questionnaire that included when the patient returned to work or school, whether a recurrence occurred, when it happened, and how it was treated. Residual postoperative chest pain was evaluated on a pain score from 0 to 5, where 0 is pain free; 1 is occasional discomfort; 2 is occasional use of analgesics; 3 is using nonopiate analgesics; 4 is regular pain using opiates; 5 is severe and intractable pain. All patients were followed for at least 12 months. Patients can come back to the clinic or visit emergency department whenever they have chest pain, dyspnea, or any signs related to the recurrence of pneumothorax.

Postoperative pulmonary function analysis Postoperative pulmonary function tests were performed for patients able to attend a hospital outpatient appointment at least 6 months after surgery. Forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1.0) were measured using a spirometer of Microspiro HI-298 (Chest Corporation, Tokyo, Japan) with the patients seated. A minimum of three acceptable forced expiratory maneuvers were performed and the best one was selected for analysis.

Data collection and statistical analysis The clinical data, operative findings, operation time, durations of postoperative chest drainage, length of hospital stay, complications, requested doses of meperidine, and data of VAS were collected.

A sample size of 446 patients (223 in each group) was originally assumed to reach clinical significance (at the .05 level with a power of 0.8) if minocycline reduced the recurrence rate from 9.8% to 2.9%.18 A planned interim analysis was conducted in March 2005 after enrollment of 200 patients with at least 12 months of follow-up. Statistical analysis was performed on an intent-to-treat basis rather than in an actual treatment basis. This study was terminated earlier than expected because the interim analysis showed a significant reduced rate of recurrence in patients receiving minocycline pleurodesis.

Continuous variables such as age or weight were expressed as the mean + standard deviation and analyzed by the two sample t-test. Categorical variables such as gender or smoking status were presented by frequency (%) and analyzed by the Fisher's exact test. Intensity of postoperative pain measured by VAS (from 0 to 10) were summarized by mean (95 percent confidence interval) and compared by Wilcoxon rank-sum test. Scores of residual chest pain were analyzed by the Wilcoxon rank-sum test. Freedom from recurrence was analyzed by the Kaplan-Meier method, and comparisons were made by the log-rank test. To identify other factors associated with recurrence of pneumothorax, the Cox regression model analyses for age (<25 vs ≧25), sex (male vs female), smoking status (yes vs no), operation indication (ipsilateral recurrence vs others), operation method (needlescopic vs conventional VATS), number of blebs (1 or 2 vs 0 or ≧3), number of endoscopic stapler cartridge, meperidine usage (yes vs no), dose of requested meperidine, and the presence of complications (yes vs no) were performed. A p value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring VATS caused by recurrent, persistent, or contralateral spontaneous pneumothorax as well as by spontaneous hemopneumothorax were eligible for this study.

Exclusion Criteria:

* greater than 50 years of age, with underlying pulmonary disease, previous ipsilateral thoracic operation, allergy to tetracycline or minocycline, and unwilling to receive randomization.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2001-06; Study Completion 2005-03

PRIMARY OUTCOMES:
The primary end point was rates of ipsilateral recurrence after the operation.

SECONDARY OUTCOMES:
safety of minocycline
early postoperative results of minocycline
long-term complication of minocycline
long-term effect on pulmonary function of minocycline pleurodesis

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — Natinal Taiwan University Hospital
Locations (1):
- Yung-Chie Lee, Taipei, Taiwan